CLINICAL TRIAL: NCT07228715
Title: A Study on a New Indicator for Assessing the Difficulty of Colonoscopy Insertion and Its Related Factors
Status: Active, not recruiting | Type: Observational
Sponsor: Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 2024467
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: the Difficulty of Colonoscopy Insertion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Junior Doctor Group
- Senior Doctor Group

SUMMARY:
This study will include adult patients undergoing painless colonoscopy at our hospital. The time required for endoscope insertion to reach the cecum (Cecal Intubation Time, CIT) by physicians of different experience levels will be recorded. CIT roughly reflects the difficulty of colonoscope insertion, which holds important clinical significance and is associated with factors such as abdominal pain, bloating, and the degree of intestinal adhesion. However, due to confounding factors such as operator experience and equipment variability, the objectivity of CIT as an indicator of insertion difficulty is reduced.

In this study, all patients' CIT data will be standardized using three different methods: Z-score standardization, median standardization, and quantile normalization. The goal is to determine which standardized form of CIT can more objectively reflect insertion difficulty and its correlation with important clinical indicators.

The purpose of this study is to establish a novel indicator that can objectively assess colonoscope insertion difficulty across different operating environments, thereby providing a scientific basis for the development of clinical treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who voluntarily undergo colonoscopy

Exclusion Criteria:

* patients who failed to complete the colonoscopy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo colonoscopy at the Second Hospital of Jilin University
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Time Required for Insertion to the Cecum (Cecal Intubation Time, CIT) | From enrollment to the end of treatment at 1 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastroenterology and Digestive Endoscopy Center, The Second Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No
Protect patients' privacy

REFERENCES:
- [Result] Dincer B, Omeroglu S, Guven O, Akgun IE, Celayir MF, Gurbulak EK, Yazici P, Koksal HM, Demir U. Factors predict prolonged colonoscopy before the procedure: prospective registry study. Surg Endosc. 2024 Oct;38(10):5704-5711. doi: 10.1007/s00464-024-11075-4. Epub 2024 Aug 13. PMID 39138684
- [Result] Lai EJ, Calderwood AH, Doros G, Fix OK, Jacobson BC. The Boston bowel preparation scale: a valid and reliable instrument for colonoscopy-oriented research. Gastrointest Endosc. 2009 Mar;69(3 Pt 2):620-5. doi: 10.1016/j.gie.2008.05.057. Epub 2009 Jan 10. PMID 19136102

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-11-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT07228715/Prot_SAP_000.pdf